CLINICAL TRIAL: NCT03953131
Title: A Pilot Study of 68Ga-Dotatate PET CT for Radiation Treatment Response Assessment in Meningiomas
Brief Title: Gallium Ga 68-DOTATATE PET/CT in Predicting Tumor Growth in Patients With Meningiomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0659; NCI-2019-00214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0659 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-05-16 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Ga(III)-DOTATOC; gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (gallium Ga 68-DOTATATE PET/CT) (Experimental): Patients receive gallium Ga 68-DOTATATE IV over a few minutes and, after 60 minutes, undergo a PET/CT scan over 5-10 minutes 14 days before starting scheduled radiation therapy and 6 weeks after completion of radiation treatment.
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga 68-DOTATATE; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Gallium Ga 68-DOTATATE — Given IV
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTATATE; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies how well gallium Ga 68-DOTATATE positron emission tomography (PET)/computed tomography (CT) works in predicting tumor growth in patients with meningiomas. Giving Gallium Ga 68-DOTATATE before PET/CT scan may work better in predicting tumor growth in patients with meningiomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of imaging with gallium Ga 68-DOTATATE (68Ga-DOTATATE) positron emission tomography/computed tomography (PET/CT).

II. To assess a metabolic response to radiation therapy in meningiomas as measured by a reduction in the tumor to background ratio of the maximum standardized uptake values (SUV) of the tumor compared to background brain parenchyma.

OUTLINE:

Patients receive gallium Ga 68-DOTATATE intravenously (IV) over a few minutes and, after 60 minutes, undergo a PET/CT scan over 5-10 minutes 14 days before starting scheduled radiation therapy and 6 weeks after completion of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any meningioma with at least 10 mm measurable residual disease.
* Age 18 years or older.
* Planned radiation therapy for meningioma.
* Ability to understand and the willingness to sign a IRB approved written informed consent document in accordance with regulatory and institutional guidelines before study entry.
* No restriction based on language that would prohibit enrollment of the participant. IRB approved VTPS form will be utilized when non-English Speaking patient is enrolled

Exclusion Criteria:

* Neurofibromatosis type 1 or 2.
* Children.
* Pregnant.
* Contraindication to MR imaging.
* Body weight greater than 400 lbs (181.4kg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Imaging with Gallium Ga 68-DOTATATE | Up to 1 year
  Lesions will be defined based on areas of T1 post contrast enhancement as assessed by magnetic resonance imaging (MRI). The largest bidimension measurements of the lesion on post-contrast T1 weighted magnetic resonance (MR) imaging will be recorded. Regions of interest (ROI) analysis of these regions of abnormal enhancement will be used to assess the max standard uptake values (SUV) of the lesion (tumor) as well as adjacent normal appearing brain parenchyma (background). These calculations will be repeated on the post-treatment scan as well as calculations for tumor to background (T/B) ratios.
Metabolic response to radiation therapy | Up to 1 year
  Will be measured by a reduction in the tumor to background ratio of the maximum SUV of the tumor compared to background brain parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org